CLINICAL TRIAL: NCT04671628
Title: Effects of a 2-week Relaxing Music Intervention on Anxiety, Stress, and Gut Symptoms in Aerobic Exercisers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Associate Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1690558
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal System--Abnormalities; Anxiety; Visceral Pain
MeSH Terms: conditions — Anxiety Disorders; Visceral Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxing music (Experimental)
  Interventions: Behavioral: Relaxing music
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Relaxing music — Participants will be asked to listen to relaxing music for 30 minutes each day. They will allowed to choose between several playlists based on their preference.
  Arms: Relaxing music

SUMMARY:
The objective of the study is to determine the impacts of a 2-week relaxing music intervention on stress, anxiety, and gut symptoms in individuals who regularly perform structured aerobic exercise. Gut symptoms like bloating, reflux, cramping, nausea, etc. are relatively common during prolonged aerobic exercise. In addition, previous research has established that levels of anxiety and stress are associated with a higher occurrence of these gut symptoms. Relaxing music has reduced anxiety in certain populations, but currently, no studies are available on its effects on anxiety, stress, and gut symptoms in people who regularly do aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* do 120+ minutes per week of planned/structured aerobic exercise of at least moderate intensity
* have had at least mild anxiety over the past 2 weeks (GAD-7 score of 5 or more)
* not currently on a psychotropic medication, or if they are on one, they must have been on a stable dose for the past three months
* not currently listening to music for relaxation purposes regularly (>60 minutes per week)
* have at least sometimes experienced gut symptoms (nausea, gas, bloating, cramping, side stitching, urge to defecate, etc.) during aerobic exercise sessions over the last month
* have access to the internet

Exclusion Criteria:

* not at least 18 years of age
* don't do 120+ minutes per week of planned/structured aerobic exercise of at least moderate intensity
* haven't had at least mild anxiety over the past 2 weeks (GAD-7 score of 5 or more)
* have recently started taking a psychotropic medication (within past 3 months)
* currently listening to music for relaxation purposes regularly (>60 minutes per week)
* have never or rarely experienced gut symptoms (nausea, gas, bloating, cramping, side stitching, urge to defecate, etc.) during aerobic exercise sessions over the last month
* don't have internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal symptom severity | The intervention will last 2 weeks. Gastrointestinal symptoms will be collected for a 1-week period before the intervention and during the 2nd week of the intervention
  The severity of several gastrointestinal symptoms will be assessed on a validated 0-10 scale.
Change in anxiety levels | The intervention will last 2 weeks. The General Anxiety Disorder-7 will be assessed before the intervention begins and again after 2 weeks.
  Levels of anxiety will be assessed with the General Anxiety Disorder-7 questionnaire. Scores on the General Anxiety Disorder-7 range from 0 to 21, with higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Change in visceral sensitivity | The intervention will last 2 weeks. The Visceral Sensitivity Index will be assessed before the intervention begins and again after 2 weeks.
  Perceptions of visceral sensitivity will be assessed via the Visceral Sensitivity Index. Scores on the Visceral Sensitivity Index can range from 0 to 75, with higher scores indicating a higher level of visceral sensitivity.
Change in perceived stress | The intervention will last 2 weeks. The Perceived Stress Scale 14 will be assessed before the intervention begins and again after 2 weeks.
  Perceived life stress will be evaluated with the Perceived Stress Scale 14. Scores on this scale can range from 0 to 56, will higher scores indicating greater amounts of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided